CLINICAL TRIAL: NCT05221489
Title: The Effects of Listening to Lullabies and Self-selected Music at Home on Prenatal Stress and Anxiety in Nulliparous Pregnant Women: A Randomized-controlled Study
Brief Title: The Effects of Listening to Lullabies and Self-selected Music on Prenatal Stress and Anxiety in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Firat University (Other)
Responsible Party: Principal Investigator, Nazlı Baltacı, Assistant Professor, phD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 368
Record Dates: First submitted 2022-01-13; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Anxiety, Stress-Related, in Pregnancy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lullaby group (Experimental): For two weeks and 30 minutes every day at home, the lullaby group (LG) only listened to the lullaby record selected by the researcher.
  Interventions: Other: listening to lullabies or self-selected music
- mix music group (Experimental): For two weeks and 30 minutes every day at home, the multi-music group (MG) listened to self-selected music from different records presented to them by the researcher.
  Interventions: Other: listening to lullabies or self-selected music
- control group (No Intervention): The control group (CG) only received routine care.

INTERVENTIONS:
Other: listening to lullabies or self-selected music — listening to lullabies for lullaby group and listening to music of their choice among various music for mix music group
  Arms: lullaby group; mix music group

SUMMARY:
Nulliparous women experience more anxiety and stress during their first transition to motherhood during pregnancy due to inexperience. The aim of this study is to compare the effects of listening to lullabies and the music of their choice at home on reducing the anxiety and stress experienced by nulliparous pregnant women.

This parallel randomized controlled trial was conducted in the obstetrics and gynecology outpatient clinics of a university hospital in eastern Turkey. Lullaby group (LG) recorded only the lullaby chosen by the researcher at home for 30 minutes a day for 2 weeks; mix music group (MG) listened to any of the music recordings presented to them by the researcher. The control group (CG) received general care only. Antenatal stress and anxiety levels were evaluated at the beginning and end of the study.

DETAILED DESCRIPTION:
Especially, nulliparous women who have experienced their first pregnancy may lose their control while making the first transition to motherhood and incorporating motherhood roles into other areas of their lives due to inexperience, and may be more vulnerable to stress and anxiety. It has been reported that these pregnant women have higher anxiety than those who have given birth. Antenatal anxiety and stress negatively affect maternal and fetal health. Health care professionals can benefit from music interventions to evaluate the anxiety and stress levels of pregnant women, especially in the last trimester, and to improve their physical, emotional and mental health. In some studies, music interventions made at home for pregnant women reduced anxiety and stress, thus providing psychological benefits during pregnancy, childbirth and postpartum period. The aim of this study is to compare the effects of listening to lullabies and the music of their choice at home on reducing the anxiety and stress experienced by nulliparous pregnant women.

This research is a randomized controlled experimental study in parallel group pretest-posttest design. The research was carried out in the obstetrics and gynecology outpatient clinics of a university hospital in eastern Turkey.

The population of the study consisted of healthy pregnant women who applied to the obstetrics clinic of the hospital where the study was conducted for pregnancy follow-up. G ∗ Power 3.1.9 software was used to calculate the sample size of the study. In the power analysis based on state and trait anxiety inventory scores, at least 35 pregnant women were included in each group with 95% confidence interval (1-α), 95.5% test power (1-β), 0.05 error and d=0.887 effect size. needed was determined. The pregnant women (n=16) included in the study were randomly assigned to the lullaby group (NG) (n=40), mixed music group (MG) (n=40) or control group (CG) (n=40) by simple randomization method. The statistician randomized the participants to intervention groups or control groups with the computer program "Quickcalcs graph pad" (http://www.graphpad.com/quickcalcs/, Accessed: 28.07.2021). Participants were grouped according to the randomization list according to the order of admission to the obstetrics clinic.

Necessary information about the study was given to the pregnant women who were suitable and willing to participate in the study. These pregnant women were randomly assigned to one of three groups after taking their written consent. There were two experimental and one control group in the study. One of the experimental group was a lullaby group and the other was a mixed music group. The control group did not listen to music, did not receive any intervention, received routine general care only during hospital visits.

First of all, sociodemographic and obstetric data of the pregnant women were collected, and their anxiety and stress levels were evaluated at the beginning of the study (pretest) and after 2 weeks of music intervention/general care (posttest). These data were collected at the hospital when pregnant women came to their pregnancy follow-ups.

Music initiatives (lullaby group and mixed music group):

The pregnant women in the lullaby group were told to listen only to the lullaby recording chosen by the researcher for 30 minutes a day for 2 weeks at home. Various music recordings consisting of "nature sounds, classical western music, Turkish music and lullaby" recordings prepared by the researchers were sent to the Mixed music group, and they were told to choose and listen to any of these recordings for 30 minutes a day for 2 weeks. Consultancy was received from a lecturer in the Musicology department regarding these music recordings. The music recordings were sent to the pregnant women through the mobile communication application (telegram, whatsapp, etc.) so that they could listen to them on their own phones, and they were asked to download/save the music recordings on their phones.

All pregnant women who were going to have a music attempt were informed about the way and conditions of listening to music at home. Based on previous studies, a guide to listening to music at home during pregnancy was developed. Accordingly, lullabies and other musical genres mentioned were used, with a slow rhythm (ranging between 60-70 beats per minute when measured with a metronome) and soft melody compatible with the normal heart rate. It was reported that pregnant women should use their own headphones in a quiet and poorly lit room to avoid being affected by ambient sounds while listening to music, they should prefer and adjust the volume of the music before listening, empty their bladder and not be hungry. The situation of performing these music attempts at home was followed up by the researcher by talking to the pregnant women on the phone every day. Researchers and participants were not blinded to the study due to the nature of the music enterprise. During the study, the routine care and follow-up of the pregnant women was not interfered with.

The data on the sociodemographic and obstetric characteristics of the pregnant women were collected with the personal information form created by the researchers in line with the literature. Anxiety and antenatal stress, which are the primary results of the study, were evaluated with the "State-Trait Anxiety Inventory" and the "Perceived Prenatal Stress Scale".

Data were evaluated using the IBM SPSS v.23 (IBM Corp. Armonk, NY, USA) program. Data were presented with descriptive statistics such as number, percentage, arithmetic mean, standard deviation. Chi-square test was used for categorical variables, and One way variance analysis (ANOVA) for the continuous variables to confirm differences in sociodemographic and obstetrics characteristics between the groups. The scores of the STAI and APSI between groups were compared using One way variance analysis (ANOVA) and Tukey test, for comparison within groups was used Paired samples t-test. Statistical significance value was accepted as p<0.05.

This study has some limitations and difficulties. The first of these; Since it is a single-center study, its results cannot be generalized to all healthy pregnant women. Latter; The long-term effectiveness of lullabies or other music concerts cannot be evaluated, since no follow-up was made during the pregnancy and postpartum period after the music attempt in the study. Third; The fact that pregnant women are asked to listen to music at home and that it is followed by phone makes it difficult to fully implement the intervention in terms of duration and conditions.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Healthy
* 19 years and older
* 36th and above gestational week
* Nulliparous
* No fetal anomaly
* Literate
* Pregnant women who have a WhatsApp application on their phone and can use this application
* Do not have a psychiatric problem
* Speaking Turkish

Exclusion Criteria:

* Unwilling to participate
* Having a risky pregnancy
* Below the 36th gestational week
* Multiparous
* Fetal anomaly
* Mental, cognitive, psychiatric, hearing and vision problems
* Illiterate
* Do not have WhatsApp application on their phone and cannot use this application
* Do not speak Turkish

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Anxiety change at 2 weeks | At baseline and at the end of the 2nd week of study, anxiety was assessed.
  As assessed by the State-Trait Anxiety Inventory
Prenatal stress change at 2 weeks | At baseline and at the end of the 2nd week of study, prenatal stress was assessed.
  As assessed by the antenatal perceived stress inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat University, Gynecology and Obstetrics Polyclinics, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author (N.B. or Ö.D.Y.) upon reasonable request.